CLINICAL TRIAL: NCT02959853
Title: Aromatase Inhibitors and Weight Loss in Severely Obese Hypogonadal Male Veterans (Pilot)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Rui Chen, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-36912
Record Dates: First submitted 2016-11-03; First posted 2016-11-09 (Estimated); Results first posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Hypogonadism; Severe Obesity
Keywords: Hypogonadism; Severe obesity
MeSH Terms: conditions — Hypogonadism; Obesity, Morbid | interventions — Anastrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- weight loss (Placebo Comparator): Patients given counseling on diet and exercise in order to achieve a goal weight loss of 10 percent
  Interventions: Behavioral: weight loss
- aromatase inhibitor (anastrazole) plus weight loss (Experimental): Patient placed on an aromatase inhibitor anastrazole 1 mg daily plus given counseling on diet and exercise in order to achieve a goal weight loss of 10 percent
  Interventions: Drug: Anastrazole; Behavioral: weight loss

INTERVENTIONS:
Drug: Anastrazole
  Other Names: Arimidex
  Arms: aromatase inhibitor (anastrazole) plus weight loss
Behavioral: weight loss

SUMMARY:
After the age of 40, there is a gradual decline in the production of testosterone. Among obese men, the decline in testosterone levels is exacerbated by the suppression of the hypothalamic-pituitary-gonadal axis by hyperestrogenemia. The high expression of aromatase enzyme in the adipose tissue enhances the conversion of androgens into estrogens which in turn exert a negative feedback on the hypothalamus and pituitary, leading to the inhibition of production of gonadotropin-releasing hormone (GnRH), luteinizing hormone (LH) and follicle stimulating hormone (FSH), and as a consequence, of testosterone by the testis resulting in hypogonadotropic hypogonadism (HH). Though bone loss is a well recognized side effect of AI in certain populations, such as women with breast cancer, HH obese men present high levels of circulating estrogens that could potentially prevent them from bone loss, estradiol being the main regulator of the male skeleton. This study is designed to determine if aromatase inhibitors in combination with weight loss, compared to weight loss alone, will have a positive effect on muscle strength, symptoms of hypogonadism, and body composition without negatively impacting bone mineral density and bone quality. Results from this study will help determine if certain groups of obese patients would benefit from therapy with aromatase inhibitors.

DETAILED DESCRIPTION:
After the age of 40, testosterone (T) production in men gradually decreases at a rate of 1.6% per year for total and to 2-3% per year for bioavailable T. Because of the age-related increase in sex hormone binding globulin, the magnitude of the decrease in bioavailable T in men is even greater than the decline in total T levels. This reduction in T production in men parallels the age-associated loss of muscle mass that leads to sarcopenia and impairment of function and the age-associated loss of bone mass that leads to osteopenia and fracture risk. Hypogonadism is a condition associated with multiple symptom complex including fatigue, depressed mood, osteoporosis, increased fat mass, loss of libido and reduced muscle strength, all of which deeply affect patient's quality of life. The prevalence of hypogonadismamong obese men ranges between 29.3% to 78.8%, with levels of androgens decreasing proportionately to the degree of obesity. This decline in T levels is exacerbated among obese patients due the suppression of the hypothalamic-pituitary-gonadal axis by hyperestrogenemia. The high expression of aromatase enzyme in the adipose tissue enhances the conversion of androgens into estrogens (E) which in turn exerts a negative feedback on hypothalamus and pituitary, inhibiting the production of gonadotropin-releasing hormone (GnRH), luteinizing hormone (LH) and follicle stimulating hormone (FSH) and, as a consequence, of T by the testis resulting in hypogonadotropic hypogonadism (HH). Considering the high aromatase expression in the adipose tissue, the administration of T among obese men with HH could increase the conversion of the substrate T to estradiol (E2) and fuels the negative feedback on the hypothalamus and pituitary, producing a greater suppression of GnRH and gonadotropins.

Thus, men with obesity induced HH may benefit from other treatment strategies that target the pathophysiology of the disease. Weight loss intervention which improves hormonal and metabolic abnormalities related to obesity may also be considered a logical approach to improve obesity-induced HH.

One possible approach consists of the use of aromatase inhibitors (AI) to stop the conversion of T to E2 thereby interrupting the vicious cycle of E2 inhibition of the hypothalamic-pituitary-gonadal axis and restoring T production to normal levels. Increased T and reduced E2 levels have been reported in men with low levels of T after AI administration, even though very few studies investigated clinical outcomes.

We believe that AI use could promote positive changes on hypogonadal symptoms and body composition in HH severely obese patients, acting at the physiopathology of the disease without necessarily causing bone loss.

ELIGIBILITY:
Inclusion Criteria:

* severely obese (BMI >= 35) male veterans with hypogonadotropic hypogonadism defined as low total testosterone (lower than 300 ng/dl) between 35-65 years of age
* Luteinizing hormone (LH) lower than 9 U/L
* estradiol above 40 pmol/l
* normal Free T4 (FT4), Thyroid Stimulating Hormone (TSH), prolactin, cortisol, Adrenocorticotropic hormone (ACTH), and Insulin-like growth factor-1 (IGF-1) levels.
* Subjects must be ambulatory, willing and able to provide written informed consent

Exclusion Criteria:

* clinical or biochemical evidence of pituitary or hypothalamic disease
* any ongoing illness that, in the opinion of the investigator, could prevent the subject from completing study
* any med known to affect gonadal hormones, steroid hormone-binding globulin or bone metabolism, e.g.,

  * androgens
  * estrogens
  * glucocorticoids
  * phenytoin
  * bisphosphonates
  * any medication known to interfere with anastrozole metabolism, e.g. tamoxifen or estrogens
* diseases known to interfere with bone metabolism as

  * osteoporosis
  * hyperparathyroidism
  * untreated hyperthyroidism
  * osteomalacia
  * chronic liver disease
  * renal failure
  * hypercortisolism
  * malabsorption
  * immobilization
  * patients with a Total T score lower than -2.0 at Lumbar Spine or Left Femur.
* patients with symptomatic prostate disease, prostate carcinoma, or elevated serum Prostate-specific antigen (PSA) >4 ng/ml or >3 for subjects with a family history of prostate cancer among 1st degree relatives needs urologic evaluation before admission into study
* hematocrit greater than 50%
* untreated severe obstructive sleep apnea
* severe lower urinary tract symptoms with International Prostate Symptom Score (IPSS) above 19
* documented heart failure
* cardiovascular disease
* liver disease
* excessive alcohol or substance abuse
* unstable weight (changes in weight more than ± 2 kg) during the last 3 months
* history of bariatric surgery
* subjects with elevated liver enzymes as alanine transaminase (ALT), aspartate aminotransferase (AST), Alkaline phosphatase (ALP), and bilirubin at greater than twice the upper limit of normal.

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reina Villareal, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas, United States

REFERENCES:
- [Derived] Colleluori G, Chen R, Turin CG, Vigevano F, Qualls C, Johnson B, Mediwala S, Villareal DT, Armamento-Villareal R. Aromatase Inhibitors Plus Weight Loss Improves the Hormonal Profile of Obese Hypogonadal Men Without Causing Major Side Effects. Front Endocrinol (Lausanne). 2020 May 15;11:277. doi: 10.3389/fendo.2020.00277. eCollection 2020. PMID 32499757

RESULTS

PARTICIPANT FLOW:
Groups:
- Weight Loss Plus Placebo: Patients given counseling on diet and exercise in order to achieve a goal weight loss of 10 percent
  weight loss
- Aromatase Inhibitor (Anastrazole) Plus Weight Loss: Patient placed on an aromatase inhibitor anastrazole 1 mg daily plus given counseling on diet and exercise in order to achieve a goal weight loss of 10 percent
  Anastrazole
  weight loss
Period: Overall Study
Arm/Group | Weight Loss Plus Placebo | Aromatase Inhibitor (Anastrazole) Plus Weight Loss
Started | 11 | 12
Completed | 7 | 10
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Population: 11 in the placebo plus weight loss group 12 in the aromatase inhibitor plus weight loss group
Groups:
- Placebo Plus Weight Loss: Patients given a placebo and counseling on diet and exercise in order to achieve a goal weight loss of 10 percent.
- Total: Total of all reporting groups
Arm/Group | Placebo Plus Weight Loss | Aromatase Inhibitor (Anastrazole) Plus Weight Loss | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 23
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 11 | 12 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 4 | 7 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Muscle Strength as Assessed by Knee Extension and Knee Flexion
Description: Muscle strength was assessed using Biodex System 4 Isokinetic Dynamometer (Shirley, NY). Peak torque for isokinetic knee extension and flexion was measured at baseline, 6 months on the right leg. During the testing, participants sat with their hips flexed at 120 degrees, secured with thigh and pelvic straps. Testing was performed at an angular velocity of 60 degrees per second. The best result of 3 maximal voluntary efforts for each knee flexion and extension was used as the measure of absolute strength and reported as peak torque at 60 degrees in Newton-meter (N*m) units.
  The higher the measured Newton-meter (N*m), the greater the measured muscle strength.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: Percent change in muscle strength
Groups:
- Weight Loss: Patients given counseling on diet and exercise in order to achieve a goal weight loss of 10 percent
  weight loss
Arm/Group | Weight Loss | Aromatase Inhibitor (Anastrazole) Plus Weight Loss
Number analyzed (Participants) | 7 | 10
Percent change in muscle strength
  percent change in knee flexion | 12.6 (13.3) | 8.9 (21.6)
  percent change in knee extension | 12.8 (13.8) | 3.7 (14.7)

2. Primary Outcome: Change in Symptoms Score of Hypogonadism
Description: Symptoms of androgen deficiency were measured with 3 validated questionnaires done at baseline, 3 and 6 months.
  1. The Quantitative Androgen Deficiency in the Aging Male (qADAM) questionnaire uses questions from a scale of 1-5. The final summation yields a total score between 10 (most symptomatic) and 50 (least symptomatic).
  2. The second questionnaire used was the International Index of Erectile Function (IIEF). Total score ranges from 5 to 25, with 5 being severe erectile dysfunction and 25 being no erectile dysfunction.
  3. The third questionnaire used was the Impact of Weight on Quality of Life Questionnaire-Lite (IWQOL-lite). Total score ranges from 31 to 155, with 31 being least symptomatic and 155 being the most symptomatic.
  Score change at 3 months calculated by: total score at 3 months minus total score at baseline
  Score change at 6 months calculated by: total score at 6 months minus total score at baseline
Time Frame: baseline, 3 and 6 months
Measure: Mean (Standard Deviation); unit: score on scale (qADAM, IIEF, IWQOL-lite)
Arm/Group | Weight Loss | Aromatase Inhibitor (Anastrazole) Plus Weight Loss
Number analyzed (Participants) | 7 | 10
score on scale (qADAM, IIEF, IWQOL-lite)
  qADAM score change at 3 months | 2.4 (3.4) | 5.8 (6.1)
  qADAM score change at 6 months | 4.1 (5.7) | 4.4 (7.2)
  IIEF score change at 3 monthss | 4.3 (3.8) | 2.7 (4.6)
  IIEF score change at 6 months | 0.9 (4.11) | 1.7 (5.8)
  IWQOL-lite score change at 3 month | -12.2 (23.9) | -13.0 (15.2)
  IWQOL-lite score change at 6 month | -16.6 (27.1) | -18.6 (8.8)

3. Secondary Outcome: Change in Fat Mass (in Kilograms)
Description: change in fat was measured by Dual-energy X-ray absorptiometry (DXA) scan at baseline and 6 months only.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Weight Loss Plus Placebo | Aromatase Inhibitor (Anastrazole) Plus Weight Loss
Number analyzed (Participants) | 7 | 10
kilograms | -0.7 (1.9) | -4.4 (3.9)

4. Secondary Outcome: Change in Visceral Adipose Tissue (in Grams)
Description: Change in absolute visceral adipose tissue as measured by DXA scan, done at baseline and 6 months.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Weight Loss Plus Placebo | Aromatase Inhibitor (Anastrazole) Plus Weight Loss
Number analyzed (Participants) | 7 | 10
grams | 28.9 (81.6) | -111.7 (258.5)

5. Secondary Outcome: Percent Change in Bone Mineral Density
Description: Percent change in bone mineral density as measured by DXA scan, done at baseline and 6 months
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Weight Loss Plus Placebo | Aromatase Inhibitor (Anastrazole) Plus Weight Loss
Number analyzed (Participants) | 7 | 10
percent change
  percent change in total hip bone density | -1.45 (3.98) | -0.46 (2.66)
  percent change in femoral neck bone density | -1.63 (2.92) | 0.82 (3.83)
  percent change in lumbar spine bone density | 3.22 (4.89) | -0.71 (3.42)

6. Secondary Outcome: Percent Change in Bone Quality
Description: Percent change in bone quality as measured by high resolution peripheral quantitative computed tomography scan (HR-pQCT), at baseline and 6 months
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Weight Loss Plus Placebo | Aromatase Inhibitor (Anastrazole) Plus Weight Loss
Number analyzed (Participants) | 7 | 5
percent change
  percent change in failure load at the radius | -2.16 (3.09) | -4.63 (6.83)
  percent change in bone stiffness at the radius | -2.09 (3.29) | -4.02 (6.42)
  percent change in failure load at the tibia | 0.80 (2.9) | -0.81 (4.62)
  percent change in bone stiffness at the tibia | 0.36 (3.28) | -1.31 (5.17)

ADVERSE EVENTS:
Time Frame: 2 years
Description: see data tables
Arm/Group | Weight Loss | Aromatase Inhibitor (Anastrazole) Plus Weight Loss
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/11 | 1/12
Other Adverse Events (participants affected / at risk) | 3/11 | 4/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weight Loss (N=11) | Aromatase Inhibitor (Anastrazole) Plus Weight Loss (N=12)
Hospital admission (Psychiatric disorders) | 1 (1) | 0 (0) — 034 admitted for suicidal ideation
Hospital (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Admitted for low back pain
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weight Loss (N=11) | Aromatase Inhibitor (Anastrazole) Plus Weight Loss (N=12)
Hot flashes (Endocrine disorders) | 0 (0) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
skin rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
heel pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
uncontrolled DM (Endocrine disorders) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/53/NCT02959853/Prot_SAP_000.pdf